CLINICAL TRIAL: NCT05818605
Title: The EXerCise traIning To rEcovery in HCM Trial
Brief Title: Exercise Intolerance in Non-obstructive Hypertrophic Cardiomyopathy
Acronym: EXCITE-HCM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL157238 (NIH); R01HL157238 (NIH)
Record Dates: First submitted 2023-04-05; First posted 2023-04-19 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, blinded
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Intensity Exercise arm (Experimental): All patients randomized to the exercise training group will undergo a single supervised in-hospital exercise session that includes an exercise consultation with a certified exercise physiologist. Following that they will exercise at-home with video supervision 3 times a week for a period of 24 weeks.
  Interventions: Behavioral: Moderate Intensity Exercise Program
- Usual physical activity arm (No Intervention): Patients randomized to the usual-activity group will be instructed to continue their current activity without initiating or intensifying any existing exercise regimens for the duration of the study

INTERVENTIONS:
Behavioral: Moderate Intensity Exercise Program — Subjects randomized to the EXER arm will undergo 24 weeks of Moderate Intensity Exercise Training (MIET). Patients will be signed up for 60-minute exercise sessions, 3 times a week
  Arms: Moderate Intensity Exercise arm

SUMMARY:
The EXCITE-HCM study is a randomized, controlled, blinded clinical trial designed to evaluate the effect of moderate intensity exercise training versus usual physicial activity on the improvement of HCM-related symptoms and cardiac function. About 70 participants will be recruited and randomized on a 1:1 ratio to either moderate intensity training or usual physicial activity interventions. Patients will be followed during a period of 24 weeks and assesesments as physical examination, questionnaires, 12 lead ecg's, biomarker levels, echocardiogram, Cardiac Magnetic resonance, PET and CPET will be performed to evaluate their response to the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 to 80 years of age with diagnosis of hypertrophic cardiomyopathy1 defined by left ventricular hypertrophy with end-diastolic wall thickness 15 mm or greater on 2D echocardiography in the absence of other primary causes of left ventricular hypertrophy or wall thickness between 13 and 15 mm in the presence of other features suggestive of hypertrophic cardiomyopathy, such as systolic anterior motion of the mitral valve leaflets, family history of hypertrophic cardiomyopathy, or positive genetic test result.
2. Left ventricular outflow tract gradient <30 mmHg at rest and with provocation.
3. Left ventricular ejection fraction ≥ 50% by biplane Simpson's method.
4. Access to exercise equipment at home or at a fitness center.
5. Ability to complete study related testing including online surveys and smart phone use
6. Ability to perform 24 weeks of exercise training

Exclusion Criteria:

1. History of exercise-induced syncope or ventricular arrhythmias
2. LVOT obstruction being evaluated for septal reduction therapy; less than 3 months after
3. History of septal reduction therapy - surgery or ablation
4. History of ICD placement in the previous 3 months
5. History of hypotensive response with exercise testing (>20 mm Hg decrease of systolic blood pressure from baseline blood pressure or an initial increase in systolic blood pressure followed by a decrease of systolic blood pressure >20 mm Hg)
6. Clinical decompensation in the previous 3 months, defined as New York Heart Association class IV congestive heart failure symptoms or Canadian Cardiovascular Society class IV angina symptoms
7. Left ventricular ejection fraction less than 50% by echocardiography
8. Life expectancy less than 12 months
9. Pregnant or planned pregnancy
10. Inability to exercise owing to any medical or other limitations
11. Unwillingness to refrain from competitive sports, burst activity, or heavy isometric exercise for the duration of the study, if assigned to the non-exercise group.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in V O2 max | Baseline and 24 weeks
  Change in peak oxygen consumption (V O2 max: mL/kg/min) by CPET
Change in peak VO2 % | Baseline and 24 weeks
  Change in peak VO2 % predicted (%) by CPET

SECONDARY OUTCOMES:
Change in Myocardial Systolic Strain | Baseline and 24 Weeks
  Change in Myocardial systolic strain (%) by echocardiography
Change in Myocardial Work | Baseline and 24 weeks
  Change Myocardial work (mmHg%) by echocardiography

OTHER OUTCOMES:
Change in Myocardial Perfussion | Baseline and 24 Weeks
  Change in Regional myocardial perfusion (ml/min/gm) by PET
Change in Coronary Flow reserve | Baseline and 24 Weeks
  Change in coronary flow reserve (ratio, no unit) by PET

CONTACTS AND LOCATIONS:
Overall Officials: Theodore P Abraham, M.D, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California - San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No